CLINICAL TRIAL: NCT01586962
Title: An Open Label, In-use Study to Assess the Warming Sensation, Acceptability and Local Tolerability of Paracetamol 500 mg + Pseudoephedrine 30 mg Syrup Given as a 30 ml Single Dose in Subjects Suffering From Symptoms of an Upper Respiratory Tract Infection
Brief Title: Warming Sensation Intensity and Acceptability of the Flavour, Local Tolerability of Paracetamol 500 mg + Pseudoephedrine 30 mg Syrup in Patients Suffering a URTI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Consumer Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 147-A-301
Record Dates: First submitted 2012-04-23; First posted 2012-04-27 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-04

CONDITIONS: Upper Respiratory Infections
Keywords: paracetamol; pseudoephedrine; syrup; upper respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Acetaminophen; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Upper Respiratory Infections (Experimental)
  Interventions: Drug: IFF flavor 316 282, Paracetamol, Pseudoephedrine

INTERVENTIONS:
Drug: IFF flavor 316 282, Paracetamol, Pseudoephedrine — Single dose syrup containing a warmingflavor IFF 316282 in a syrup containing Paracetamol and pseudoephedrine

SUMMARY:
This is an open label, in-use study to assess the warming sensation, acceptability and local tolerability of paracetamol 500 mg + pseudoephedrine 30 mg syrup, given as a single dose in subjects suffering from symptoms of an upper respiratory tract infection. The purpose is to evaluate the acceptability concerning a warming sensation effect and its potential benefit in the target population.

The primary objective is to assess the warming sensation caused by the excipient IFF flavor 316 282, in a syrup containing paracetamol 500 mg + pseudoephedrine 30 mg per 30 ml syrup. The syrup contains (0.15% w/v) warming flavor.

The Secondary Objectives are to assess subject acceptability of the syrup and the safety and tolerability of the syrup. The study will be run in fifty-six (56) subjects suffering from symptoms of an upper respiratory tract infection (URTI) for 7 days or less, e.g. nasal congestion associated with colds and flu symptoms such as pain, headache and/or fever. Subjects must have one or more symptoms per category:

1. mild to moderate body pain, headache, fever or sore throat
2. nasal congestion (blocked nose) with or without rhinorrhea (runny nose) or sneezing Adolescents will be included in the study population

ELIGIBILITY:
Inclusion Criteria:

* Subject must have one or more symptoms per category (see also screening assessment of cold symptoms, section 6.1):
* mild to moderate body pain, headache, fever or sore throat
* nasal congestion (blocked nose) with or without rhinorrhea (runny nose) or sneezing

Exclusion Criteria:

1. Baseline sore throat pain of severe intensity, e.g. rated as 3 on a 4-point ordinal scale (0=not present, 1= mild, 2=moderate, 3=severe)
2. Baseline dry cough of severe intensity, e.g. rated as 3 on a 4-point ordinal scale (0=not present, 1= mild, 2=moderate, 3=severe)
3. Subject has a productive cough.
4. History of hypersensitivity to any of the study drugs and the listed excipients or to drugs of similar chemical classes
5. Subjects with allergic asthma.
6. Use of any inhaler, medicated confectionary, throat lozenges, throat pastilles, sprays, any products with demulcent properties such as chewing gums and boiled sweets or mints, in the 6 hours prior to dosing.
7. Use of any medication for sore throat containing a local anaesthetic within the 6 hours prior to dosing.
8. Use of paracetamol, any NSAID or any oral nasal decongestant within 6 hours prior to dosing.
9. Use of substances of abuse or antihistamines within 24 hours of dosing.
10. Drinking of tea, coffee or other caffeinated beverages 1 hour prior to dosing.
11. Suffering from hepatic or severe renal impairment, hypertension, hyperthyroidism, diabetes, heart disease or other acute or chronic medical condition that, in the opinion of the investigator, would put the subject at a higher risk or affect the conduct and/or the results of the study.
12. Use of any antidepressants, monoamine oxidase inhibitors or beta-blocking drugs in the 28 days prior to dosing
13. A history of alcohol abuse or subject admits to regular consumption of alcohol in excess of the recommended weekly limits of 21 units for females and 28 units for males.
14. Subject is a current smoker of ≥10 cigarettes per day (or reports equivalent smoking habits using other tobacco products).
15. Subject has smoked or chewed tobacco products within 12 hours of dosing.
16. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Algorithme Pharma, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start/End Dates 07 May 2012 to 17 May 2012
Groups:
- Upper Respiratory Infections: IFF flavor 316 282, Paracetamol, Pseudoephedrine : Single dose syrup containing a warmingflavor IFF 316282 in a syrup containing Paracetamol and pseudoephedrine
Period: Overall Study
Arm/Group | Upper Respiratory Infections
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Upper Respiratory Infections
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.8 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 25
Region of Enrollment [Number; unit: participants]
  Canada | 56

OUTCOME MEASURES:

1. Primary Outcome: Warming Sensation Caused by the Excipient IFF Flavor 316 282, in a Syrup Containing Paracetamol 500 mg + Pseudoephedrine 30 mg Per 30 ml Syrup
Description: Intensity of warming sensation felt by subjects between predose to 1 minute postdose where 0 = no warming sensation and 100 = strongest possible warming sensation
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Upper Respiratory Infections
Number analyzed (Participants) | 56
mm | 34.2 (25.51)

2. Secondary Outcome: Subject Acceptability of the Syrup
Description: How do you like the warming sensation you have experienced for this product?
  Possible responses are :
  Like extremely Like very much Like moderately Like slightly Neither like nor dislike Dislike slightly Dislike moderately Dislike very much Dislike extremely
Time Frame: 1 hour
Measure: Number; unit: Participants
Arm/Group | Upper Respiratory Infections
Number analyzed (Participants) | 56
Participants | 39

3. Secondary Outcome: Safety and Tolerability of the Syrup
Description: Number of participants with adverse events.
Time Frame: 1 hour
Measure: Number; unit: Participants
Arm/Group | Upper Respiratory Infections
Number analyzed (Participants) | 56
Participants | 9

ADVERSE EVENTS:
Arm/Group | Upper Respiratory Infections
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 4/56
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Upper Respiratory Infections (N=56)
Somnolence (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator